CLINICAL TRIAL: NCT06610149
Title: A Multicenter Real-World, Single-Arm, Open-Label Study Assessing the Impact of Novel Probiotic Mixture on the Symptoms of Irritable Bowel Syndrome in Adults
Brief Title: A Novel Probiotic Mixture in Adults With IBS
Acronym: IBS-dammil5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Prof, University of Bari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PENTA-IBS
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Single-Arm, Open-Label Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): 8-week treatment period with a probiotic mixture (Lactobacillus paracasei 101/37 LMG P-17504, Lactobacillus plantarum 14D CECT 4528, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve BL10 LMG P-17500, and Bifidobacterium animalis ssp. lactis Bi1 LMG P-17502)
  Interventions: Dietary Supplement: Probiotic mixture

INTERVENTIONS:
Dietary Supplement: Probiotic mixture — 8 weeks treatment with Probiotic mixture

SUMMARY:
Irritable bowel syndrome (IBS) is faced by gastroenterologists on a daily basis and probiotics are a potential therapeutic tool, however, there is no strain recommendations. This multicenter re-al-world, single-arm, open-label study aims to assess the effectiveness, safety, and patient satis-faction of a novel probiotic mixture in patients with IBS. Methods: This study is conducted by Italian gastroenterologists who enroll patients with IBS. Throughout the 8-week treatment (T1) period with a probiotic mixture (Lactobacillus paracasei 101/37 LMG P-17504, Lac-tobacillus plantarum 14D CECT 4528, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve BL10 LMG P-17500, and Bifidobacterium animalis ssp. lactis Bi1 LMG P-17502), participants complete a questionnaire to evaluate IBS symptoms at baseline, at the end of treatment, and after one-month follow-up (T2).

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is faced by gastroenterologists on a daily basis and probiotics are a potential therapeutic tool, however, there is no strain recommendations. This multicenter re-al-world, single-arm, open-label study aims to assess the effectiveness, safety, and patient satis-faction of a novel probiotic mixture in patients with IBS. Methods: This study is conducted by Italian gastroenterologists who enroll patients with IBS. Throughout the 8-week treatment (T1) period with a probiotic mixture (Lactobacillus paracasei 101/37 LMG P-17504, Lac-tobacillus plantarum 14D CECT 4528, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve BL10 LMG P-17500, and Bifidobacterium animalis ssp. lactis Bi1 LMG P-17502), participants complete a questionnaire to evaluate IBS symptoms at baseline, at the end of treatment, and after one-month follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* recurrent abdominal pain at least once per week during the past three months associated with two or more of the following criteria:
* related to defecation,
* Associated with a change in the frequency of stool,
* Associated with a change in the appearance of stool.

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1098 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
abdominal pain | After 8 weeks of probiotic supplementation and after 4 weeks of follow-up
  abdominal pain severity. The questionnaire utilized a 5-point Likert scale, where 0 represented the absence of symptoms, and 5 indicated the presence of highly intense symptoms. Treatment success will be defined as a change towards categories of lower IBS severity for abdominal pain and/or bloating 149 between inclusion (T0) and the end of the supplementation period (T1)
bloating | After 8 weeks of probiotic supplementation and after 4 weeks of follow-up
  bloating severity. The questionnaire utilized a 5-point Likert scale, where 0 represented the absence of symptoms, and 5 indicated the presence of highly intense symptoms. Treatment success will be defined as a change towards categories of lower IBS severity for abdominal pain and/or bloating 149 between inclusion (T0) and the end of the supplementation period (T1).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Pediatrica, Bari, Apulia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drago L, Corleto VD, Ciprandi G, Brindicci VF, Dargenio VN, Cristofori F, Schettini F, Mauro A, Di Marino VP, la Grasta G, Marseglia G; IBSdammil5 study group; Francavilla R. A multicenter real-world, open-label study assessing the impact of a probiotic mixture on symptoms of irritable bowel syndrome in adults. Benef Microbes. 2025 Sep 16:1-12. doi: 10.1163/18762891-bja00097. Online ahead of print. PMID 40987448